CLINICAL TRIAL: NCT00959829
Title: Use of Music and Vocal Stimulus in Patients in Coma State - Relations Between Auditory Stimulus, Vital Signs, Face Expression and Glasgow Coma Scale or Ramsay Scale
Brief Title: Use of Music and Voice Stimulus on Coma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Ana Claudia Giesbrecht Puggina, Escola de Enfermagem da Universidade de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FAPESP 03/10035-4
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2009-08

CONDITIONS: Coma
Keywords: Communication; Complementary Therapies; Intensive Care; Ethics
MeSH Terms: conditions — Coma; Communication

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- silence (Placebo Comparator): The control group listened "silence" and was evaluated the same things.
  Interventions: Other: Music and message

INTERVENTIONS:
Other: Music and message — Experimental group: music and message Control group: silence
  Other Names: Patients in state of coma or induced coma

SUMMARY:
Objectives: (1) To check music and voice message influence on vital signs and facial expressions of patients in physiological or induced comas; (2) To connect the existence of patient's responsiveness with the Glasgow Coma Scale or with the Ramsay Sedation Scale.

Method: This was a randomized controlled clinical trial with 30 patients, from two Intensive Care Units, being divided in 2 groups (control and experimental). Their relatives recorded a voice message and chose a song according to the patient's preference. The patients were submitted to 3 sessions for 3 consecutive days.

DETAILED DESCRIPTION:
The relatives elaborated a voice recorded message and choose a music according to the patient preference, which were recorded in the same Compact Disc. Two identical CD's were made at the same recorded time; one with and another one without stimulus in order to make the random division of the groups. The patients were evaluated according to one of the Scales; they used earphones. During the sessions, the data relating to the vital signs and the face expression were recorded in a data collection instrument.

ELIGIBILITY:
Inclusion Criteria:

* To be in coma;
* To be evaluated according to one of the Scales and to have a score in the study range: in physiological comas, score between 3 to 8 Glasgow Coma Scale (GCS); in induced coma, one of the last two scores of Ramsay Sedation Scale (RSS), R5 or R6;
* To have hearing function preserved according to family;
* To have written consent from the family or responsible party for the patient's participation in the research.

Exclusion Criteria:

* Score between 9 to 15 in GCS or scores R1, R2, R3 or R4 in RSS

Ages: 16 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-02; Primary Completion 2005-03 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Vital signs | 3 days; before and after stimulus or silence

CONTACTS AND LOCATIONS:
Locations (1):
- HCFMUSP - Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Puggina AC, Silva MJ. [Vital signs and facial expression of patients in coma]. Rev Bras Enferm. 2009 May-Jun;62(3):435-41. doi: 10.1590/s0034-71672009000300016. Portuguese. PMID 19597668